CLINICAL TRIAL: NCT06520865
Title: Identification and Validation of a Biomarker for Tinnitus: an Objective Data-driven Personalized Approach to Diagnosis of Chronic Tinnitus - The Tinnitus Detection (TIDE) Project
Brief Title: TIDE Project: Biomarker Discovery for Chronic Tinnitus Diagnosis
Acronym: TIDE
Status: Completed | Type: Observational
Sponsor: University of Regensburg (Other)
Collaborators: University of Dublin, Trinity College (Other); Universität Tübingen (Other); University Hospital, Zürich (Other); Eastern Switzerland University of Applied Sciences (Other); University of Texas at Austin (Other); University of Illinois at Urbana-Champaign (Other); Brain - Brain Research Center for Advanced, Innovative, Interdisciplinary and International Neuromodulation (Unknown)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., Prof. Dr. med., University of Regensburg
Other Study IDs: TIDE
Record Dates: First submitted 2024-07-22; First posted 2024-07-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Tinnitus
Keywords: Tinnitus, Biomarker for Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tinnitus cases/patients: Subjects that have a diagnosis of chronic and constant tinnitus (for at least 6 months based on history)
  Interventions: Other: Acoustic paradigms
- Control group: Subjects that never experienced tinnitus (excluding short-term tinnitus, i.e. not tinnitus that persists over a longer period of time)
  Interventions: Other: Acoustic paradigms

INTERVENTIONS:
Other: Acoustic paradigms — Acoustic oddball Gap detection

SUMMARY:
Research in clinical neuroscience is founded on the conviction that a better understanding of tinnitus related changes of brain function will improve our ability to diagnose and treat tinnitus. Although considerable advances have been made in understanding the mechanisms of tinnitus, the clinical management of tinnitus remains largely based on a 'trial and error' approach. The identification and validation of a biomarker for tinnitus is thought to be the crucial step in the development of a personalized approach to the diagnosis and treatment of tinnitus. The overarching goal of this study is to incorporate advanced technologies to provide an objective, data-driven, personalized approach to the diagnosis of chronic tinnitus. This should lead to a clinically applicable tool that can be widely and easily used.

DETAILED DESCRIPTION:
The tinnitus detect (TIDE) consortium has been designed to identify and validate a biomarker for the presence and intensity of tinnitus. For this purpose, two test paradigms are combined which are derived from the most recent models of tinnitus and which have shown promise in pilot studies.

A first approach is based on a method used in animals to objectively assess tinnitus by gap detection, namely Gap prepulse inhibition of the acoustic startle (GPIAS). The GPIAS paradigm is inspired from the combination of both gap detection and pre-pulse inhibition (PPI), used for the assessment of temporal sensory processing in both animals and humans. The basic principle of PPI relies on the ability of a weak lead stimulus (a prepulse or a silent gap presented in a carrier background) to inhibit a startling effect of a following, more intense, abrupt stimulus. These paradigms have been used to assess the automatic or preconscious inhibition of the motor reflex response that occurs in healthy subjects. Because GPIAS is regulated at the level of the auditory cortex, cortical responses may provide a more accurate measure of inhibition than motor reflex responses, such as the startle response in animals or the eye blinking in humans. The hypothesis is that individuals with tinnitus would have impaired inhibition of cortical evoked responses to sound pulses when preceded by a silent gap, in comparison to non-tinnitus individuals, due to the ongoing tinnitus percept.

A second approach is based on the concept that tinnitus occurrence is related to altered processing of prediction errors. This concept is supported by empirical evidence demonstrating that people with tinnitus exhibit a more pronounced electrophysiological response to a mismatch between predictions (the expected sound based on the auditory training paradigm) and perceptions as compared to non-tinnitus individuals. This sensitivity to prediction errors (the difference between prediction and input) is associated with how loud patients perceive their tinnitus, independent of co-occurring hyperacusis and hearing loss. For example, the amplitude of the mismatch negativity (MMN) positively correlates with subjectively reported tinnitus loudness. Thus, the MMN might be a biomarker for how loud tinnitus patients perceive their tinnitus. That is, people with a more pronounced electrophysiological response to a prediction error perceive a louder phantom sound. Using another paradigm, a group, independent of us, confirmed the importance of the MMN for tinnitus detection. Furthermore, an increase in amplitude and a delay in latency for the late positive evoked brain response (P300) has been demonstrated in tinnitus patients using both auditory and visual oddball paradigms. Both the MMN and P300 are conceived as measures of prediction errors identified at respectively the sensory cortex and higher levels (i.e., frontal-parietal cortex). The P300 is thought to reflect processes involved in stimulus evaluation or categorization; whether the stimulus is behaviourally relevant or not. Therefore, the aim of the current approach is to validate that both the MMN and the P300, using an auditory oddball paradigm with omission, can be used as biomarkers for tinnitus loudness and presence, respectively, (i.e., cross-validation).

We propose to investigate these two paradigms in a large international sample of tinnitus patients and controls in order to determine the sensitivity of GPIAS and the oddball paradigm in diagnosing tinnitus in humans.

ELIGIBILITY:
Inclusion Criteria:

(1) for tinnitus cases: a diagnosis of chronic and constant tinnitus (for at least 6 months based on history)

* (2) for controls: never experienced tinnitus
* (3) age 18 -70;
* (4) ability to understand and consent to the research;
* (5) ability to participate (hearing ability);
* (6) MoCa Test ≥ 26;
* (7) hyperacusis questionnaire score < 27;
* (8) Hospital Anxiety and Depression Scale (HADS) <14;

Exclusion Criteria:

* (1) objective tinnitus; heartbeat-synchronous tinnitus as primary complaint;
* (2) otosclerosis; acoustic neuroma or other relevant ear disorders with fluctuating hearing;
* (3) acute ear nose and throat infections (acute otitis media, otitis externa, acute sinusitis);
* (4) Meniere's disease or similar syndromes;
* (5) vestibular migraine;
* (6) serious internal, neurological or psychiatric conditions;
* (7) epilepsy or other CNS disorders (brain tumor, encephalitis);
* (8) clinically relevant drug, medication or alcohol abuse up to 12 weeks before study start;
* (9) change in anti-depressants/drugs ≤ 2 weeks
* (10) missing written informed consent
* (11) severe hearing loss - inability to communicate properly in the course of the study;
* (12) one deaf ear;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with chronic tinnitus (for at least 6 months) and control subjects who have never had (except short-term) tinnitus.
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Event-related potentials | 4 hours
  Event-related potentials of a 64-channel EEG

CONTACTS AND LOCATIONS:
Overall Officials: Sven Vanneste, Prof., Principal Investigator — Trinnitus College Dublin
Locations (7):
- United States (2):
  - University of Illinois, Champaign, Illinois
  - University of Texas, Austin, Texas
- Brai3n - Research center for Advanced, International, Innovative and Interdisciplinary Neuromodulation, Ghent, Belgium
- Germany (2):
  - University of Tuebingen, Tübingen, Baden-Wurttemberg
  - Center of Neuromodulation - Psychiatry und Psychotherapie der Universität Regensburg am Bezirksklinikum, Regensburg, Bavaria
- Trinity College Dublin, Dublin, Ireland
- OST - Eastern Switzerland University of Applied Sciences, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided